CLINICAL TRIAL: NCT01546649
Title: A Phase 3 Comparative Study of TAP-144-SR(6M) in Postoperative and Hormone Therapy-naïve Patients With Premenopausal Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP-144-SR(6M)IP/CPH-202; JapicCTI-121762 (Registry Identifier: JapicCTI); U1111-1128-7039 (Registry Identifier: WHO)
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Premenopausal Breast Cancer

ARMS (2):
- TAP-144-SR(6M) (Experimental): TAP-144-SR(6M) 22.5 mg, injection, treatment interval 24 weeks for up to 96 weeks.
  Interventions: Drug: TAP-144-SR(6M)
- TAP-144-SR(3M) (Active Comparator): TAP-144-SR(3M) 11.25 mg, injection, treatment interval 12 weeks for up to 96 weeks.
  Interventions: Drug: TAP-144-SR(3M)

INTERVENTIONS:
Drug: TAP-144-SR(6M)
  Arms: TAP-144-SR(6M)
Drug: TAP-144-SR(3M)
  Arms: TAP-144-SR(3M)

SUMMARY:
Hormone dynamics, pharmacokinetics, safety, and efficacy of TAP-144-SR(6M) will be evaluated against TAP-144-SR(3M) in postoperative and hormone therapy-naïve patients with premenopausal breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. The participant has histopathologically-confirmed primary breast cancer in Japanese.
2. The participant is aged 20 years or older when informed consent is obtained
3. The participant has estrogen receptor (ER)-positive tumor cells and/or progesterone receptor (PgR)-positive primary tumor. And HER-2 is negative.
4. The participant has breast cancer in the clinical stages of T1-T3, N-any and M0 by TNM classification (the seventh edition, proposed by UICC in 2009). (No distant metastasis to lung, liver and bone should be confirmed on the image-based diagnosis at study enrollment. The image taken within 12 weeks prior to study enrollment is also available for the diagnosis.) The number of axillary lymph node metastasis is not limited.
5. Any operative procedure for breast cancer is acceptable. In principle, after breast-conserving surgery, the participant will receive postoperative radiation to the conserving breast.
6. Neoadjuvant chemotherapy and adjuvant chemotherapy prior to study enrollment are acceptable. (It is advisable the same kind of chemotherapy is performed at each site.)
7. The participant has a history of regular menstrual periods within 12 weeks prior to study enrollment, or the participant has FSH of less than 40 mIU/mL and E2 of 10 pg/mL or more measured within 12 weeks prior to study enrollment. The participant has not had a chemical menopause (i.e., FSH of less than 40 mIU/mL and E2 of 10 pg/mL or more) within 12 weeks after completing adjuvant chemotherapy.
8. The participant is in a condition to receive study drug and Tamoxifen (TAM) within 12 weeks after surgery or after adjuvant chemotherapy prior to study enrollment. Adjuvant chemotherapy prior to study is required to have been completed at the time of study enrollment.
9. The participant has ECOG performance status of grades 0 or 1 at the time of study enrollment.
10. The participant meets the following criteria of hepatic, renal and bone marrow functions on the laboratory test results at screening:

    * Hepatic function: AST (GOT) ≤ 3.0 times the upper limit of normal (ULN) ALT (GPT) ≤ 3.0 times the ULN
    * Renal function: serum creatinine level < 1.5 times the ULN
    * Bone marrow function : white blood cell count ≥ 3,000/mm3 platelet count ≥ 100,000/μL hemoglobin ≥ 10.0g/dL
11. The participant agrees to use a non-hormonal method of contraception through the study period.

Exclusion Criteria:

1. The participant has received neoadjuvant or adjuvant hormonal therapy for the latest breast cancer surgery.
2. The participant has received bilateral oophorectomy and bilateral ovarian irradiation.
3. The participant has inflammatory breast cancer or bilateral breast cancer.
4. The participant has non-invasive ductal carcinoma.
5. The participant has multiple primary cancers, or a history of carcinoma in other organs.
6. The participant is pregnant or breast-feeding.
7. The participant has a history of hypersensitivity to synthetic LH-RH, LH-RH derivative, TAM, TAM analogue (antiestrogen) or any component of the study drug.
8. The participant has a history of, or has been diagnosed with thromboembolism including myocardial infarction, cerebral infarction, venous thrombosis, and pulmonary embolism, or cardiac failure.
9. Patients whose QTcF interval exceeded 460 msec on the 12-lead electrocardiogram at screening.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Nagoya, Aichi-ken
  - Fukushima, Fukushima
  - Maebashi, Gunma
  - Ohta-shi, Gunma
  - Sapporo, Hokkaido
  - Isehara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Nigata-shi, Niigata
  - Kurashiki-shi, Okayama-ken
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Kita-adachi-gun, Saitama
  - Shinjuku-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 21 investigative sites in Japan from April 2012 to December 2014.
Pre-assignment Details: Participants with a historical diagnosis of premenopausal breast cancer were enrolled in 1 of 2 treatment groups as follows: TAP-144-SR(6M); TAP-144-SR(3M)
Groups:
- TAP-144-SR (6M): TAP-144-SR (6M) 22.5 milligram (mg), injection, subcutaneous, once in 24 weeks along with tamoxifen 20 mg, tablet, orally, once daily for up to 96 weeks.
- TAP-144-SR (3M): TAP-144-SR (3M) 11.25 mg, injection, subcutaneous, once in 12 weeks along with tamoxifen 20 mg, tablet, orally, once daily for up to 96 weeks.
Period: Overall Study
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Started | 83 | 84
Completed | 75 | 75
Not Completed | 8 | 9
Not completed — Adverse Event | 4 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Recurrence | 1 | 1
Not completed — Discovery of secondary cancer | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who had received at least a single dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M) | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (4.90) | 44.0 (5.18) | 44.1 (5.03)
Age, Customized [Number; unit: participants]
  Less than (<) 40 years | 13 | 12 | 25
  Greater than equal to (>=) 40 to <45 years | 29 | 30 | 59
  >=45 years | 41 | 42 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 84 | 167
  Male | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 159.3 (5.11) | 158.1 (5.00) | 158.7 (5.08)
Height, Customized [Number; unit: participants]
  <150 cm | 2 | 3 | 5
  >=150 to <160 cm | 40 | 53 | 93
  >=160 cm | 41 | 28 | 69
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 54.48 (7.670) | 53.57 (7.498) | 54.02 (7.574)
Weight, Customized [Number; unit: participants]
  <50 kg | 25 | 29 | 54
  >=50 to <60 kg | 40 | 40 | 80
  >=60 kg | 18 | 15 | 33
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.50 (3.042) | 21.45 (2.902) | 21.48 (2.964)
BMI, Customized [Number; unit: participants]
  <18.5 kg/m^2 | 8 | 13 | 21
  >=18.5 to <25.0 kg/m^2 | 63 | 61 | 124
  >=25.0 to <30.0 kg/m^2 | 12 | 9 | 21
  >=30.0 kg/m^2 | 0 | 1 | 1
Surgical procedure, Customized [Number; unit: participants]
  Breast-conserving surgery | 53 | 58 | 111
  Mastectomy | 30 | 26 | 56
Pathological diagnosis, Customized [Number; unit: participants]
  Papillotubular carcinoma | 33 | 36 | 69
  Solid-tubular carcinoma | 7 | 4 | 11
  Scirrhous carcinoma | 30 | 34 | 64
  Mucinous carcinoma | 4 | 1 | 5
  Invasive lobular carcinoma | 6 | 6 | 12
  Tubular adenocarcinoma | 1 | 0 | 1
  Invasive micropapillary carcinoma | 1 | 3 | 4
  Specified neoplasms (other) | 1 | 0 | 1
TNM classification: clinical tumor stage T, Customized [Number; unit: participants] — The frequency of clinical tumor stage T (0, 1, 2, 3, 4, X, or Tis) was assessed. The frequency of T was evaluated prior to surgery. The categories of T are ranged from 0 (No evidence of primary tumor) to 4 (Tumor of any size with direct extension to chest wall and/or to skin). X is representing tumor cannot be evaluated, 0 is representing no signs of tumor, Tis is carcinoma in situ.
  participants
    T1 | 63 | 64 | 127
    T2 | 19 | 18 | 37
    T3 | 1 | 2 | 3
TNM classification: regional lymph node stage N, Customized [Number; unit: participants] — The frequency of regional lymph nodes stage N (0, 1, 2, 3, or X) was assessed. The frequency of N was evaluated prior to surgery. The categories of N are ranged from 0 (No regional lymph node metastasis) to 3 (Metastasis in ipsilateral infraclavicular lymph node(s); or in clinically detected ipsilateral internal mammary lymph node(s); or metastasis in ipsilateral supraclavicular lymph node(s)). X is representing lymph nodes cannot be evaluated, 0 is tumor cells absent from regional lymph nodes.
  participants
    N0 | 78 | 81 | 159
    N1 | 5 | 3 | 8
TNM classification: M0 [Number; unit: participants] — The frequency of distant metastasis clinical stage M (0, 1) was assessed. The frequency of M was evaluated prior to surgery. The categories of M are represented by 0 (no distant metastasis) and 1 (distant metastasis).
  participants | 83 | 84 | 167
TNM staging (Stage), Customized [Number; unit: participants] — The stage of cancer based on TNM classification: Stage 0 (Carcinoma in situ which is staged by Tis, N0, M0), Stage IA (T1, N0, M0), IB (T0/T1, N1, M0), IIA (T0/T1, N1, M0 or T2, N0, M0), IIB (T2, N1, M0 or T3, N0, M0), IIIA (T0/T1/T2, N2, M0 or T3, N1/N2, M0), IIIB (T4, N0/N1/N2, M0) and IIIC (Any T, N3, M0), Stage IV(Any T, Any N, M1).
  participants
    I | 61 | 61 | 122
    IIA | 19 | 21 | 40
    IIB | 2 | 2 | 4
    IIIA | 1 | 0 | 1
Histopathological tumor size [Mean (Standard Deviation); unit: cm] | 1.64 (1.312) | 1.55 (1.023) | 1.59 (1.173)
Histopathological tumor size, Customized [Number; unit: participants]
  Less than equal to (<=) 2.0 cm | 65 | 66 | 131
  >2.0 cm | 18 | 18 | 36
Axillary lymph node metastases [Mean (Standard Deviation); unit: number of metastases] | 0.2 (0.46) | 0.2 (0.57) | 0.2 (0.52)
Axillary lymph node metastases, Customized [Number; unit: participants]
  Present | 15 | 14 | 29
  Absent | 68 | 70 | 138
Axillary lymph node metastases, Customized [Number; unit: participants]
  0 | 68 | 70 | 138
  >=1 metastasis to <=3 metastases | 15 | 14 | 29
  >=4 metastases | 0 | 0 | 0
Time from surgery or previous postoperative adjuvant therapy to administration of study drug [Number; unit: participants]
  <=28 days | 6 | 9 | 15
  >=29 to <=56 days | 42 | 43 | 85
  >=57 days | 35 | 32 | 67
Primary tumor estrogen receptors (ER)/ progesterone receptors (PgR) status, Customized [Number; unit: participants]
  ER -positive / PgR-positive | 82 | 82 | 164
  ER -positive / PgR -negative | 1 | 2 | 3
  ER -negative / PgR -positive | 0 | 0 | 0
Human epidermal growth factor receptor 2 (HER2) (immunohistochemistry [IHC] scoring), Customized [Number; unit: participants] — Participants with HER expression by IHC was reported as 0, 1+, 2+, 3+, or unmeasured. The categories of HER expression is ranged from 0 (better) to 3+ (worse).
  participants
    0 | 37 | 33 | 70
    1+ | 33 | 28 | 61
    2+ | 7 | 13 | 20
    3+ | 0 | 0 | 0
    Not performed | 6 | 10 | 16
HER2 (fluorescent in situ hybridization [FISH] testing), Customized [Number; unit: participants]
  Positive | 0 | 0 | 0
  Negative | 13 | 23 | 36
  Equivocal | 0 | 0 | 0
  Not performed | 70 | 61 | 131
The eastern cooperative oncology group performance status (ECOG P.S.), Customized [Number; unit: participants] — Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair.
  participants
    0 | 83 | 84 | 167
    1 | 0 | 0 | 0
Menstruation (before the first dose), Customized [Number; unit: participants]
  Present | 82 | 81 | 163
  Absent | 1 | 3 | 4
Time from last menstruation to first dose [Mean (Standard Deviation); unit: days] | 17.0 (13.27) | 15.9 (14.28) | 16.4 (13.75)
Time from last menstruation to first dose, Customized [Number; unit: participants]
  <=28 days | 72 | 73 | 145
  >=29 to <=56 days | 8 | 6 | 14
  >=57 days | 2 | 2 | 4
  Missing | 1 | 3 | 4
Serum Estradiol (E2) concentration (pretreatment) [Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)] | 168.0 (162.99) | 138.2 (125.45) | 153.0 (145.66)
Serum E2 concentration (pretreatment), Customized [Number; unit: participants]
  <=29 pg/mL | 7 | 11 | 18
  >=30 pg/mL | 76 | 73 | 149
Radiation, Customized [Number; unit: participants] — Participants were classified based on whether they had received radiation therapy or not.
  participants
    Present | 52 | 59 | 111
    Absent | 31 | 25 | 56
Preoperative and postoperative chemotherapy, Customized [Number; unit: participants]
  Present | 0 | 1 | 1
  Absent | 83 | 83 | 166
Previous breast cancer (other), Customized [Number; unit: participants]
  Present | 0 | 0 | 0
  Absent | 83 | 84 | 167
Concomitant osteoporosis medication , Customized [Number; unit: participants]
  Present | 6 | 9 | 15
  Absent | 77 | 75 | 152
Smoking Classification, Customized [Number; unit: participants]
  Never Smoked | 55 | 54 | 109
  Current Smoker | 9 | 11 | 20
  Ex-smoker | 19 | 19 | 38
Time from surgery or previous postoperative adjuvant therapy to administration of study drug [Mean (Standard Deviation); unit: days] | 55.4 (21.69) | 51.8 (16.01) | 53.6 (19.08)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppressive Effect of Serum Estradiol (E2) to Menopausal Level (=<30 pg/mL) From Week 4 Through Week 48
Description: Comparison of both the treatment groups was done by assessing the suppressive effect on serum E2 concentration maintained at menopausal level (=<30pg/mL). Suppression rate was calculated as proportion of participants maintained at menopausal level.
Time Frame: Week 4 up to Week 48
Population: Full analysis set (FAS) included all randomized participants who had received at least a single dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
percentage of participants | 97.6 [91.565 to 99.707] | 96.4 [89.916 to 99.257]

2. Secondary Outcome: Concentration of Serum E2
Description: The measure indicates serum E2 concentration at baseline and post-baseline time points.
Time Frame: Baseline, Hour (hr) 1, 3, 6 on Day 1, Day 2, 3, 4, 8, 15, 22, 29, 57, 85, 113, 141, 169, 176, 183, 197, 225, 253, 281, 309, 337, 421, 505, 589 and 673
Population: FAS included all randomized participants who had received at least a single dose of study treatment. Here 'N' represents evaluable baseline and post-baseline assessment population.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
pg/mL
  Baseline [N=83;84] | 95 [0 to 652] | 99 [0 to 533]
  Day1 (1hr) [N=82;84] | 94.5 [0 to 616] | 110.5 [0 to 518]
  Day1 (3hr) [N=24;21] | 102.0 [0 to 602] | 64.0 [15 to 404]
  Day1 (6hr) [N=24;21] | 153.5 [0 to 681] | 99.0 [16 to 533]
  Day2 [N=83;84] | 146.0 [0 to 693] | 115.5 [0 to 333]
  Day3 [N=83;84] | 100.0 [0 to 417] | 87.5 [0 to 311]
  Day4 [N=83;84] | 108.0 [0 to 543] | 110.0 [0 to 453]
  Week 1 (Day8) [N=83;84] | 56.0 [0 to 904] | 112.0 [0 to 981]
  Week 2 (Day15) [N=83;84] | 13.0 [0 to 866] | 0.0 [0 to 1220]
  Week 3 (Day22) [N=83;84] | 0.0 [0 to 196] | 0.0 [0 to 722]
  Week 4 (Day29) [N=83;84] | 0.0 [0 to 14] | 0.0 [0 to 50]
  Week 8 (Day57) [N=83;84] | 0.0 [0 to 12] | 0.0 [0 to 158]
  Week 12 (Day85) [N=83;83] | 0.0 [0 to 12] | 0.0 [0 to 11]
  Week 16 (Day113) [N=82;82] | 0.0 [0 to 69] | 0.0 [0 to 16]
  Week 20 (Day141) [N=81;82] | 0.0 [0 to 15] | 0.0 [0 to 15]
  Week 24 (Day169) [N=80;81] | 0.0 [0 to 27] | 0.0 [0 to 20]
  Week 25 (Day176) [N=79;80] | 0.0 [0 to 18] | 0.0 [0 to 15]
  Week 26 (Day183) [N=79;80] | 0.0 [0 to 14] | 0.0 [0 to 19]
  Week 28 (Day197) [N=75;77] | 0.0 [0 to 14] | 0.0 [0 to 16]
  Week 32 (Day225) [N=78;80] | 0.0 [0 to 17] | 0.0 [0 to 18]
  Week 36 (Day253) [N=79;80] | 0.0 [0 to 18] | 0.0 [0 to 17]
  Week 40 (Day281) [N=78;80] | 0.0 [0 to 184] | 0.0 [0 to 12]
  Week 44 (Day309) [N=77;80] | 0.0 [0 to 16] | 0.0 [0 to 15]
  Week 48 (Day337) [N=77;80] | 0.0 [0 to 15] | 0.0 [0 to 19]
  Week 60 (Day421) [N=77;79] | 0.0 [0 to 25] | 0.0 [0 to 21]
  Week 72 (Day505) [N=77;78] | 0.0 [0 to 14] | 0.0 [0 to 18]
  Week 84 (Day589) [N=76;77] | 0.0 [0 to 15] | 0.0 [0 to 14]
  Week 96 (Day673) [N=75;75] | 0.0 [0 to 12] | 0.0 [0 to 24]

3. Secondary Outcome: Concentration of Serum Luteinizing Hormone (LH)
Description: This measure indicates serum LH concentration at baseline and post-baseline time points. It was measured in milli-international units per milliliter (mIU/mL).
Time Frame: Baseline, Hour 1, 3, 6 on Day 1, Day 2, 3, 4, 8, 15, 22, 29, 57, 85, 113, 141, 169, 176, 183, 197, 225, 253, 281, 309, 337, 421, 505, 589 and 673
Population: as for outcome 2
Measure: Median (Full Range); unit: mIU/mL
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
mIU/mL
  Baseline [N=83;84] | 4.250 [0.69 to 65.33] | 4.490 [0.77 to 40.17]
  Day1 (1hr) [N=82;84] | 27.730 [8.12 to 250.00] | 30.585 [2.78 to 207.30]
  Day1 (3hr) [N=24;21] | 88.020 [24.64 to 250.00] | 63.260 [12.00 to 153.60]
  Day1 (6hr) [N=24;21] | 64.750 [32.54 to 198.90] | 61.210 [12.68 to 106.10]
  Day2 [N=83;84] | 14.990 [3.22 to 90.63] | 19.755 [1.84 to 154.30]
  Day3 [N=83;84] | 7.310 [1.28 to 27.86] | 10.500 [1.73 to 59.52]
  Day4 [N=83;84] | 5.830 [1.13 to 41.16] | 9.375 [1.63 to 56.11]
  Week 1 (Day8) [N=83;84] | 3.190 [0.75 to 25.08] | 4.475 [1.18 to 29.68]
  Week 2 (Day15) [N=83;84] | 2.460 [0.76 to 10.56] | 1.990 [0.75 to 9.65]
  Week 3 (Day22) [N=83;84] | 1.020 [0.24 to 4.39] | 1.085 [0.38 to 5.35]
  Week 4 (Day29) [N=83;84] | 0.540 [0.16 to 1.85] | 0.845 [0.33 to 2.73]
  Week 8 (Day57) [N=83;84] | 0.270 [0.00 to 1.15] | 0.570 [0.00 to 5.17]
  Week 12 (Day85) [N=83;83] | 0.220 [0.00 to 1.84] | 0.520 [0.00 to 2.70]
  Week 16 (Day113) [N=82;82] | 0.245 [0.00 to 7.08] | 0.430 [0.00 to 1.42]
  Week 20 (Day141) [N=81;82] | 0.240 [0.00 to 2.26] | 0.405 [0.00 to 2.93]
  Week 24 (Day169) [N=80;81] | 0.290 [0.00 to 8.01] | 0.460 [0.11 to 2.96]
  Week 25 (Day176) [N=79;80] | 0.450 [0.00 to 7.92] | 0.455 [0.15 to 1.47]
  Week 26 (Day183) [N=79;80] | 0.410 [0.12 to 2.46] | 0.405 [0.14 to 1.70]
  Week 28 (Day197) [N=75;77] | 0.270 [0.11 to 0.95] | 0.410 [0.11 to 1.68]
  Week 32 (Day225) [N=78;80] | 0.280 [0.00 to 1.31] | 0.440 [0.14 to 2.45]
  Week 36 (Day253) [N=79;80] | 0.250 [0.00 to 2.02] | 0.395 [0.11 to 2.01]
  Week 40 (Day281) [N=78;80] | 0.240 [0.00 to 2.05] | 0.390 [0.12 to 1.75]
  Week 44 (Day309) [N=77;80] | 0.250 [0.00 to 2.67] | 0.385 [0.00 to 2.14]
  Week 48 (Day337) [N=77;80] | 0.250 [0.00 to 2.12] | 0.415 [0.11 to 1.30]
  Week 60 (Day421) [N=77;79] | 0.250 [0.00 to 1.52] | 0.440 [0.00 to 2.57]
  Week 72 (Day505) [N=77;78] | 0.260 [0.00 to 1.24] | 0.420 [0.00 to 1.91]
  Week 84 (Day589) [N=76;77] | 0.230 [0.00 to 1.30] | 0.410 [0.00 to 1.34]
  Week 96 (Day673) [N=75;75] | 0.210 [0.00 to 1.48] | 0.360 [0.00 to 1.63]

4. Secondary Outcome: Concentration of Follicle Stimulating Hormone (FSH)
Description: This measure indicates serum FSH concentration at baseline and post-baseline time points.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: mIU/mL
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
mIU/mL
  Baseline [N=83;84] | 5.070 [1.97 to 57.33] | 5.605 [2.03 to 66.13]
  Day1 (1hr) [N=82;84] | 9.520 [4.01 to 102.42] | 10.000 [4.02 to 99.71]
  Day1 (3hr) [N=24;21] | 23.325 [8.39 to 110.28] | 19.950 [10.06 to 74.66]
  Day1 (6hr) [N=24;21] | 27.460 [11.19 to 147.78] | 25.340 [10.85 to 107.69]
  Day2 [N=83;84] | 10.080 [2.78 to 93.70] | 12.515 [3.23 to 115.42]
  Day3 [N=83;84] | 6.180 [2.86 to 45.56] | 6.780 [3.09 to 55.25]
  Day4 [N=83;84] | 6.100 [2.84 to 37.79] | 5.585 [2.75 to 36.28]
  Week 1 (Day8) [N=83;84] | 3.920 [0.99 to 14.09] | 3.035 [1.19 to 11.62]
  Week 2 (Day15) [N=83;84] | 1.820 [0.58 to 7.49] | 1.705 [0.47 to 4.63]
  Week 3 (Day22) [N=83;84] | 1.220 [0.49 to 3.22] | 1.570 [0.49 to 4.68]
  Week 4 (Day29) [N=83;84] | 1.200 [0.39 to 2.48] | 2.015 [0.68 to 7.37]
  Week 8 (Day57) [N=83;84] | 1.390 [0.36 to 5.15] | 2.345 [0.87 to 7.75]
  Week 12 (Day85) [N=83;83] | 1.490 [0.37 to 5.72] | 2.240 [0.76 to 7.06]
  Week 16 (Day113) [N=82;82] | 1.635 [0.59 to 11.04] | 1.830 [0.69 to 4.82]
  Week 20 (Day141) [N=81;82] | 1.780 [0.53 to 7.28] | 1.905 [0.87 to 8.76]
  Week 24 (Day169) [N=80;81] | 2.060 [0.42 to 6.24] | 2.000 [0.59 to 6.52]
  Week 25 (Day176) [N=79;80] | 1.940 [0.71 to 5.22] | 1.600 [0.51 to 4.25]
  Week 26 (Day183) [N=79;80] | 1.560 [0.53 to 3.40] | 1.700 [0.64 to 3.71]
  Week 28 (Day197) [N=75;77] | 1.310 [0.52 to 2.81] | 1.690 [0.59 to 5.91]
  Week 32 (Day225) [N=78;80] | 1.595 [0.52 to 4.81] | 1.980 [0.57 to 4.69]
  Week 36 (Day253) [N=79;80] | 1.660 [0.73 to 6.12] | 2.035 [0.67 to 5.49]
  Week 40 (Day281) [N=78;80] | 1.735 [0.75 to 4.09] | 1.710 [0.71 to 7.62]
  Week 44 (Day309) [N=77;80] | 1.930 [0.72 to 5.01] | 1.825 [0.70 to 6.39]
  Week 48 (Day337) [N=77;80] | 1.920 [0.69 to 8.37] | 1.885 [0.72 to 4.09]
  Week 60 (Day421) [N=77;79] | 1.530 [0.74 to 4.71] | 1.910 [0.64 to 4.75]
  Week 72 (Day505) [N=77;78] | 1.730 [0.92 to 5.89] | 1.920 [0.63 to 4.30]
  Week 84 (Day589) [N=76;77] | 1.500 [0.77 to 3.23] | 1.840 [0.66 to 3.74]
  Week 96 (Day673) [N=75;75] | 1.620 [0.76 to 4.57] | 1.740 [0.59 to 7.01]

5. Secondary Outcome: Disease Free Survival (DFS) Rate at Week 96
Description: DFS is defined as time from randomization to earliest day of onset the events, recurrence [including recurrence in the ipsilateral breast], secondary cancer [including breast cancer in the contralateral breast] and death. DFS at Week 96 was defined as the percentage, calculated with Kaplan-Meier method, of participants did not experience any events at Week 96 since the randomization.
Time Frame: Week 96
Population: FAS included all randomized participants who had received at least a single dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
percentage of participants | 97.3 | 97.5

6. Secondary Outcome: Distant Disease Free Survival (DDFS) Rate at Week 96
Description: DDFS is defined as time from randomization to earliest day of onset the events, distant recurrence, secondary cancer [including breast cancer in the contralateral breast] and death. DDFS at week 96 was defined as the percentage calculated with Kaplan-Meier method, of participants did not experience any events at week 96 since the randomization.
Time Frame: Week 96
Population: FAS included all randomized participants who had received at least a single dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
percentage of participants | 98.5 | 98.8

7. Secondary Outcome: Serum Unchanged TAP-144 Level
Description: This measure indicates the unchanged TAP-144 level in serum.
Time Frame: Baseline, Hour 1, 3, 6 on Day 1, Day 2, 3, 4, 8, 15, 22, 29, 57, 85, 113, 141, 169, 176, 183, 197, 225, 253, 281, 309 and 337
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram per deciliter (ng/dL)
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
nanogram per deciliter (ng/dL)
  Baseline [N=83;84] | 0.000 (0.0000) [0.69 to 65.33] | 0.000 (0.0000) [0.77 to 40.17]
  Day1 (1hr) [N=82;84] | 5.293 (1.0684) [8.12 to 250.00] | 28.45 (9.7398) [2.78 to 207.30]
  Day1 (3hr) [N=24;19] | 2.538 (0.46023) [24.64 to 250.00] | 20.27 (3.9535) [12.00 to 153.60]
  Day1 (6hr) [N=24;21] | 1.039 (0.23264) [32.54 to 198.90] | 8.037 (1.7408) [12.68 to 106.10]
  Day2 [N=83;84] | 0.1401 (0.066137) [3.22 to 90.63] | 0.4749 (0.17801) [1.84 to 154.30]
  Day3 [N=83;84] | 0.02889 (0.026108) [1.28 to 27.86] | 0.2492 (0.097054) [1.73 to 59.52]
  Day4 [N=83;84] | 0.02380 (0.022645) [1.13 to 41.16] | 0.2273 (0.080794) [1.63 to 56.11]
  Week 1 (Day8) [N=82;83] | 0.09115 (0.22637) [0.75 to 25.08] | 0.1050 (0.049062) [1.18 to 29.68]
  Week 2 (Day15) [N=82;84] | 0.3702 (0.25134) [0.76 to 10.56] | 0.08867 (0.077142) [0.75 to 9.65]
  Week 3 (Day22) [N=83;84] | 0.7285 (0.35639) [0.24 to 4.39] | 0.06471 (0.092279) [0.38 to 5.35]
  Week 4 (Day29) [N=83;83] | 0.3442 (0.19814) [0.16 to 1.85] | 0.04971 (0.032917) [0.33 to 2.73]
  Week 8 (Day57) [N=83;83] | 0.1146 (0.053068) [0.00 to 1.15] | 0.04744 (0.032379) [0.00 to 5.17]
  Week 12 (Day85) [N=83;83] | 0.08051 (0.041881) [0.00 to 1.84] | 0.06028 (0.031104) [0.00 to 2.70]
  Week 16 (Day113) [N=82;82] | 0.05775 (0.037098) [0.00 to 7.08] | 0.09347 (0.077284) [0.00 to 1.42]
  Week 20 (Day141) [N=81;82] | 0.03941 (0.037082) [0.00 to 2.26] | 0.07165 (0.062739) [0.00 to 2.93]
  Week 24 (Day169) [N=80;81] | 0.02931 (0.019785) [0.00 to 8.01] | 0.07634 (0.064118) [0.11 to 2.96]
  Week 25 (Day176) [N=79;80] | 0.1128 (0.16751) [0.00 to 7.92] | 0.1583 (0.089299) [0.15 to 1.47]
  Week 26 (Day183) [N=79;80] | 0.3327 (0.36474) [0.12 to 2.46] | 0.1109 (0.065133) [0.14 to 1.70]
  Week 28 (Day197) [N=80;80] | 0.4687 (0.36083) [0.11 to 0.95] | 0.08468 (0.040820) [0.11 to 1.68]
  Week 32 (Day225) [N=78;80] | 0.1377 (0.093340) [0.00 to 1.31] | 0.06881 (0.037607) [0.14 to 2.45]
  Week 36 (Day253) [N=79;80] | 0.08521 (0.040324) [0.00 to 2.02] | 0.06259 (0.036687) [0.11 to 2.01]
  Week 40 (Day281) [N=79;80] | 0.06073 (0.032232) [0.00 to 2.05] | 0.08163 (0.031631) [0.12 to 1.75]
  Week 44 (Day309) [N=77;80] | 0.4339 (0.026552) [0.00 to 2.67] | 0.06479 (0.028540) [0.00 to 2.14]
  Week 48 (Day337) [N=77;80] | 0.02957 (0.017147) [0.00 to 2.12] | 0.06313 (0.032149) [0.11 to 1.30]

8. Secondary Outcome: QT Interval Measured by 12-lead Electrocardiogram (ECG)
Description: 12-lead electrocardiography measurement was performed in supine position after 5 minutes at rest. Each measurement was recorded continuously for 10 seconds at the recording speed of 25 millimeter/second (mm/second).
Time Frame: Baseline, Hour 1, 3, 6 on Day 1, Day 29, 85, 169 and 337
Population: Safety evaluation was conducted in the safety analysis set (SAS). Here 'N' represents evaluable baseline and post-baseline assessment population.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Number analyzed (Participants) | 83 | 84
millisecond (msec)
  Baseline [N=83;84] | 421.5 (16.05) [0.69 to 65.33] | 420.9 (16.53) [0.77 to 40.17]
  Day1 (1hr) [N=83;84] | 417.8 (15.37) [8.12 to 250.00] | 417.1 (17.83) [2.78 to 207.30]
  Day1 (3hr) [N=24;21] | 416.8 (11.34) [24.64 to 250.00] | 423.7 (18.90) [12.00 to 153.60]
  Day1 (6hr) [N=24;21] | 415.8 (18.68) [32.54 to 198.90] | 424.1 (13.76) [12.68 to 106.10]
  Week 4 (Day29) [N=83;84] | 431.2 (19.30) [0.16 to 1.85] | 432.3 (16.90) [0.33 to 2.73]
  Week 12 (Day85) [N=83;84] | 433.3 (19.44) [0.00 to 1.84] | 432.3 (20.01) [0.00 to 2.70]
  Week 24 (Day169) [N=81;82] | 431.0 (21.22) [0.00 to 8.01] | 429.0 (20.28) [0.11 to 2.96]
  Week 48 (Day337) [N=77;80] | 430.0 (17.31) [0.00 to 2.12] | 431.4 (18.89) [0.11 to 1.30]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAP-144-SR (6M) | TAP-144-SR (3M)
Serious Adverse Events (participants affected / at risk) | 6/83 | 7/84
Other Adverse Events (participants affected / at risk) | 82/83 | 82/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAP-144-SR (6M) (N=83) | TAP-144-SR (3M) (N=84)
Eyelid ptosis (Eye disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Occult blood positive (Investigations) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Behcet's syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAP-144-SR (6M) (N=83) | TAP-144-SR (3M) (N=84)
Palpitations (Cardiac disorders) | 7 | 3
Conjunctivitis (Eye disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 7 | 9
Constipation (Gastrointestinal disorders) | 13 | 2
Vomiting (Gastrointestinal disorders) | 6 | 4
Gastritis (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Toothache (Gastrointestinal disorders) | 0 | 7
Injection site induration (General disorders) | 36 | 33
Injection site pain (General disorders) | 24 | 26
Malaise (General disorders) | 13 | 13
Injection site erythema (General disorders) | 13 | 8
Injection site swelling (General disorders) | 12 | 5
Injection site bruising (General disorders) | 5 | 7
Pyrexia (General disorders) | 4 | 5
Hepatic steatosis (Hepatobiliary disorders) | 6 | 8
Nasopharyngitis (Infections and infestations) | 47 | 42
Influenza (Infections and infestations) | 8 | 4
Cystitis (Infections and infestations) | 5 | 3
Radiation skin injury (Injury, poisoning and procedural complications) | 31 | 39
Radiation pneumonitis (Injury, poisoning and procedural complications) | 7 | 3
Procedural pain (Injury, poisoning and procedural complications) | 3 | 6
Wound complication (Injury, poisoning and procedural complications) | 2 | 5
White blood cell count decreased (Investigations) | 27 | 19
Weight increased (Investigations) | 12 | 8
Gamma-glutamyltransferase increased (Investigations) | 3 | 12
Electrocardiogram QT prolonged (Investigations) | 7 | 4
Blood creatine phosphokinase increased (Investigations) | 5 | 3
Bone density decreased (Investigations) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 20
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 11 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 | 3
Headache (Nervous system disorders) | 21 | 19
Dizziness (Nervous system disorders) | 6 | 9
Somnolence (Nervous system disorders) | 0 | 6
Insomnia (Psychiatric disorders) | 10 | 9
Menopausal symptoms (Reproductive system and breast disorders) | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 7
Rash (Skin and subcutaneous tissue disorders) | 9 | 6
Eczema (Skin and subcutaneous tissue disorders) | 3 | 9
Hot flush (Vascular disorders) | 43 | 48
Hypertension (Vascular disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.